CLINICAL TRIAL: NCT06397729
Title: Evaluation of a Novel Technology to Support Tailored Health Behavior Counseling in Rural Primary Care Clinics
Acronym: Rural PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Missouri Highlands Health Care (Unknown)
Responsible Party: Principal Investigator, Maura Mohler Kepper, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202309157
Record Dates: First submitted 2024-01-23; First posted 2024-05-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Obesity
Keywords: Digital health; Behavior Change; Physical Activity; Diet; Cardiovascular Disease; Obesity; Rural health
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients - Wait-List Control (Active Comparator): * Complete questionnaires at baseline, within 48 hours of their routine clinic visit, and 6-months after the clinic visit. All surveys will be administered electronically or by mail
  * A PREVENT action plan (behavior change prescription, community resources, and education) will be provided to the patient via email after the completion of the follow-up measurement.
  Interventions: Behavioral: Wait-List Control
- Patients- PREVENT Tool (Experimental): * Complete questionnaires at baseline, within 48 hours of their routine clinic visit, and 6-months after the clinic visit. All surveys will be administered electronically or by mail
  * At the clinic visit, the provider will use the PREVENT tool to discuss CVH risk and deliver a tailored behavioral change plan inclusive of patient-centered community resources. Community Health Workers will follow up with patients monthly to support behavior change.
  Interventions: Behavioral: PREVENT Tool
- Providers (No Intervention): All eligible providers will be sent questionnaires electronically to their email at baseline, following provider training and follow-up. Providers will be invited to attend a training session to educate them on the PREVENT tool at baseline.

INTERVENTIONS:
Behavioral: Wait-List Control — Will receive routine clinical care. After completion of follow-up measures, control participants will receive a behavior change prescription via the PREVENT tool
  Arms: Patients - Wait-List Control
Behavioral: PREVENT Tool — PREVENT is a novel Health Information Technology tool designed to promote physical activity and healthy food intake among overweight/obese patients at the point of care. PREVENT automates the delivery of personalized, evidence-based behavior change recommendations and provides an interactive map of community resources to help the care team link patients to resources in their community. PREVENT follows up with patients electronically and communicates progress on behavior change to the care team.
  Arms: Patients- PREVENT Tool

SUMMARY:
This project will conduct a pilot hybrid study that examines the implementation (Aims 1 & 2) and preliminary effectiveness (Aim 3) of PREVENT, a digital health intervention, among patients with overweight/obesity (N=100) using a clinic-randomized design. The central hypothesis of the study is that PREVENT will be feasible and show improvements in health behavior counseling and the patient experience that will improve patients' motivation to change, and their CVH health behaviors and outcomes.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) prevalence is 40% higher among rural than urban residents in the United States. Maintaining healthy weight, physical activity, and food intake behaviors promotes cardiovascular health (CVH) and prevents CVD. The Health Resources and Services Administration requires health behavior counseling and follow-up care for patients with elevated body mass index. Counseling is most effective when developed with and tailored to the patient and offered with resources that support healthy food intake and physical activity. Healthcare teams are challenged by the lack of accessible evidence-based, tailored recommendations and limited awareness of patient health behaviors and community resources, all of which are compounded by lack of time within the clinical workflow. Yet, digital health tools that can facilitate quality counseling and follow-up are not readily available for primary care teams - particularly those in low-resourced rural settings. The investigators will leverage our existing digital health tool (PREVENT) for healthcare teams, including Community Health Workers (CHWs), to use at the point-of-care with rural low-income patients who are overweight or obese and often have more severe social needs. PREVENT visually displays patient-reported and electronic health record data to facilitate counseling and deliver tailored physical activity and healthy food intake goals and resources. The investigators have been working with the Missouri Highlands Health Care, a federally-qualified health center with 10 clinics across 7 rural counties that has an existing CHW network, to adapt our tool to meet the needs of their health care teams and patients. This project will examine the implementation (Aims 1 & 2) and preliminary effectiveness (Aim 3) of PREVENT among patients with overweight/obesity (N=100) using a clinic-randomized design in four clinics. The investigators believe that PREVENT will be feasible and show improvements in health behavior counseling and the patient experience that will improve patients' motivation to change, CVH health behaviors, and outcomes. The investigators will seek to understand factors impacting implementation and sustainment of this approach to streamline the translation of this tool into routine care. Our ultimate goal is to improve CVH with enhanced health behavior counseling and follow-up using a multi-level approach that targets health behaviors and unmet social needs to give everyone an equal opportunity for health.

ELIGIBILITY:
Patient Inclusion Criteria:

* Aged 18-64 years at baseline
* Low income (household income <200% FPL)
* At risk for poor CVH (body mass index greater than or equal to 30)
* Receiving care from the Missouri Highlands Healthcare
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)

Provider Inclusion Criteria:

• All providers and clinic staff (physicians, nurses, community health workers, clinic staff, clinic research associates) in the Missouri Highlands Healthcare Clinics are eligible to participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Healthcare team member confidence | baseline, at study completion (3 years)
  A survey (4-questions) will assess provider's confidence in delivering health behavior counseling and discussing cardiovascular health with patients. Questions are asked on a 5-point Likert scale (range: 4-20) with a higher score indicating greater satisfaction. Change in confidence from baseline to post-study will be compared in intervention clinics versus control clinics.
Quality counseling | Within 48 hours of clinic visit
  A 12 question survey will ask patients 1) if they have been counseled on 10 topics Life's Essential 8 (obesity, blood pressure, physical activity, food intake, smoking, sleep, cholesterol, and diabetes), and two distractor topics (flu vaccination and seat belt use); 2) if they received goals for healthy eating and/or physical activity; and 3) if they received resources to support their health. Discussion of physical activity and/or food intake will satisfy that health behavior counseling was delivered. Yes' to physical activity or food intake counseling and 'yes' to receipt of tailored goals and/or resources will satisfy the 'quality behavioral counseling' outcome.

SECONDARY OUTCOMES:
Provider satisfaction | at study completion (3 years)
  A survey (33-questions) will assess provider's acceptability and satisfaction with five aspects of health information technology (content, accuracy, format, ease of use and timeliness) and PREVENT's fit with their clinic workflow. Questions are asked on a 5-point Likert scale (range: 33-165) with a higher score indicating greater satisfaction.
Shared Decision Making | 3 months into study
  Direct observation of intervention visits will be conducted using the Observing Patient Involvement in Decision Making instrument62 to understand the extent to which the PREVENT tool facilitates shared decision making.
Resource Offering | 6-months
  The number and type of resources offered will be tracked by PREVENT for each patient
Patient satisfaction | Within 48 hours of clinic visit
  A survey (6-questions) will assess patient's satisfaction with the PREVENT tool. Questions are asked on a 5-point Likert scale (range: 6-30) with a higher score indicating greater satisfaction.
Patient motivation to change | at baseline, and 6-months
  A survey (11-question) administered to patients will assess motivation and self-efficacy for behavior change. Questions are asked using a 5-point Likert scale (range: 11-55) with a higher score indicating greater motivation.
Change in patients knowledge of CVH | at baseline, and 6-months
  A survey (4-question) administered to patients to assess their knowledge of CVH risk (perceived value/importance of healthy behaviors) and awareness of resources. Questions are asked using a 5-point Likert scale (range: 4-20) with a higher score indicating greater knowledge.
Change in food intake behaviors | at baseline, and 6-months
  Patients report servings per week or per day for fruit intake, vegetable intake, whole grains, sugar-sweetened beverages, fast food consumption, and snacking behaviors.
Change in physical activity behaviors | at baseline, and 6-months
  Patient-reported physical activity (minutes of moderate and vigorous activity per week) are collected using a survey (4-questions). Patients report the average number of minutes of moderate and vigorous activity they do per week.
Change in body mass index (BMI) index z-score | At baseline, and 6-months
  Collected from patient's medical record.
Change on patient's average systolic and diastolic blood pressure | At baseline, and 6-months
  Collected from patient's medical record
Change in patient's cholesterol at baseline and at study completion | At baseline, and 6-months
  Collected from patient's medical record
Change in patient's blood glucose at baseline and at study completion | At baseline, and 6-months
  Collected from patient's medical record

CONTACTS AND LOCATIONS:
Overall Officials: Maura Kepper, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No